CLINICAL TRIAL: NCT00180310
Title: A Clinical Evaluation of the XIENCE V® Everolimus Eluting Coronary Stent System in the Treatment of Patients With de Novo Native Coronary Artery Lesions
Brief Title: SPIRIT II: A Clinical Evaluation of the XIENCE V® Everolimus Eluting Coronary Stent System
Acronym: SPIRIT II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Kathleen Peeters, Abbott Vascular
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03-364
Record Dates: First submitted 2005-09-11; First posted 2005-09-16 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Coronary Disease; Coronary Artery Disease; Coronary Restenosis
Keywords: drug eluting stents; stents; angioplasty; coronary artery disease; total coronary occlusion; coronary artery restenosis; stent thrombosis; vascular disease; myocardial ischemia; coronary artery stenosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Coronary Restenosis; Vascular Diseases; Myocardial Ischemia; Coronary Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): XIENCE V® Everolimus Eluting Coronary Stent System
  Interventions: Device: XIENCE V® Everolimus Eluting Coronary Stent
- 2 (Active Comparator): TAXUS™ EXPRESS2™ Paclitaxel Eluting Coronary Stent
  Interventions: Device: TAXUS™ EXPRESS2™ Paclitaxel Eluting Coronary Stent

INTERVENTIONS:
Device: XIENCE V® Everolimus Eluting Coronary Stent — Drug eluting stent implantation stent in the treatment of coronary artery disease.
  Other Names: XIENCE V® Everolimus Eluting Coronary Stent System
  Arms: 1
Device: TAXUS™ EXPRESS2™ Paclitaxel Eluting Coronary Stent — Drug eluting stent implantation stent in the treatment of coronary artery disease
  Other Names: TAXUS™ EXPRESS2™ Paclitaxel Eluting Coronary Stent System
  Arms: 2

SUMMARY:
Prospective, randomized, active-control, single blind, parallel two-arm multi-center clinical trial comparing XIENCE V® Everolimus Eluting Coronary Stent System to the approved commercially available active control TAXUS™ EXPRESS2™ Paclitaxel Eluting Coronary Stent System.

TAXUS™ EXPRESS2™ Paclitaxel Eluting Coronary Stent System is manufactured by Boston Scientific.

DETAILED DESCRIPTION:
The SPIRIT II trial was a randomized, single blind, active control, multi-center clinical evaluation. Subject eligibility criteria were similar to SPIRIT III and enrollment duration overlapped between studies. In this study, 300 subjects (3:1 randomization XIENCE V® EECSS: TAXUS™ PECSS were enrolled at 31 sites outside the United States. The primary endpoint was in-stent late loss at 6 months. Secondary endpoints included clinical outcomes at months 1, 6, and 9 months and 1, 2, 3, 4 and 5 years; angiographic results at 6 months and 2 years; and IVUS results at 6 months and 2 years. Follow-up through 3 years is currently available.

ELIGIBILITY:
Inclusion Criteria:

* De novo Target lesion(s) must be located in a native epicardial vessel with diameter between 2.25 mm and 4.25 mm by visual estimate
* The target lesion(s) must be in a major artery or branch with a visually estimated stenosis of >= 50% and < 100% with a TIMI flow of >= 1
* Non-study, percutaneous intervention for lesions in a non-target vessel is allowed if done >= 90 days prior to the index procedure or if planned to be done > 9 months after the index procedure

Exclusion Criteria:

* De novo target lesion(s) located in a major epicardial vessel or a side branch that has been previously treated with any type of percutaneous intervention (e.g., balloon angioplasty, stent, cutting balloon, atherectomy) < 9 months prior to index procedure
* Target lesion(s) restenotic from previous intervention
* Target lesion(s) located in a major epicardial vessel that has been previously treated with brachytherapy
* Target vessel(s) contains visible thrombus
* Patient has a high probability that a procedure other than pre-dilatation, stenting and post-dilatation will be required at the time of index procedure for treatment of the target vessel (e.g. atherectomy, cutting balloon or brachytherapy)
* Patient has additional clinically significant lesion(s) (> 50% diameter stenosis) in a target vessel or side branch for which an intervention within 9 months after the index procedure may be required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2005-07; Primary Completion 2007-07 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
In-stent late loss (LL) | at 180 days

SECONDARY OUTCOMES:
In-segment Late Loss | at 180 days (all patients) and at 2 years (for a subset of 152 patients)
In-stent Late Loss at 2 years (for a subset of 152 patients) | at 2 years (for a subset of 152 patients)
Proximal and distal Late Loss | at 180 days (all patients) and at 2 years (for a subset of 152 patients)
In-stent and in-segment Angiographic Binary Restenosis (ABR) rate | at 180 days (all patients) and at 2 years (for a subset of 152 patients)
In-stent and in-segment percent Diameter Stenosis (% DS) | at 180 days (all patients) and at 2 years (for a subset of 152 patients)
In-stent percent Volume Obstruction (% VO) | at 180 days and at 2 years for a subset of 152 patients
Plaque behind the stent( by IVUS) | at 180 days and at 2 years for a subset of 152 patients
Ischemia Driven Major Adverse Cardiac Event (ID-MACE) rate | at 30, 180 and 270 days, 1, 2, 3, 4 and 5 years
Ischemia Driven Target Vessel Failure (ID-TVF) | at 30, 180 and 270 days, 1, 2, 3, 4 and 5 years
Ischemia Driven Target Lesion Revascularization (ID-TLR) | at 30, 180 and 270 days, 1, 2, 3, 4 and 5 years
Persisting incomplete stent apposition, late-acquired incomplete stent apposition | at 180 days and at 2 years for a subset of 152 patients
Aneurysm, thrombosis and persisting dissection | at 180 days (all patients) and at 2 years (for a subset of 152 patients)
Acute success(device, procedure and clinical) | Acute

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Serruys, Principal Investigator — Erasmus Medical Center, Thoraxcenter, Rotterdam, the Netherlands
Locations (32):
- Wilheminenspital der Stadt Wien, Vienna, Austria
- Belgium (3):
  - A.Z. Middelheim, Antwerp
  - C.H.R. La Citadelle, Liège
  - C.H.U. de Liège Sart Tilman, Liège
- Denmark (3):
  - Aalborg Sygehus Syd, Aalborg
  - Århus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
- France (5):
  - Hôpital Cochin, Paris
  - Clinique Saint Hilaire, Rouen
  - Clinique Pasteur, Toulouse
  - Hôpital de Rangueil CHU, Toulouse
  - Clinique Saint Gatien, Tours
- Germany (5):
  - Herzzentrum Bad Oeynhausen, Bad Oeynhausen
  - Segeberger Kliniken GmbH, Bad Segeberg
  - Amper Kliniken AG Klinikum Dachau, Dachau
  - Herz- und Gefäßzentrum Hamburg, Hamburg
  - Klinikum Kassel, Kassel
- Max Devki Devi Heart & Vascular Institute, New Delhi, India
- Azienda Ospedaliera Santa Maria Nuova, Reggio Emilia, Italy
- Netherlands (5):
  - Academisch Medisch Centrum, Amsterdam
  - Amphia Hospital, Breda
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
  - Erasmus Medical Center, Rotterdam
  - Isala Klinieken - Locatie Weezenlanden, Zwolle
- New Zealand (2):
  - The Mercy Hospital, Auckland, Epsom
  - Auckland City Hospital, Auckland, Grafton
- National Institute of Cardiology in Warsaw, Warsaw, Poland
- Vergelegen Mediclinic, Cape Town, South Africa
- Spain (2):
  - Hospital Clinico San Carlos, Madrid
  - University Hospital Gregorio Maranon, Madrid
- Switzerland (2):
  - Kantonsspital Basel, Basel
  - R.V. Hôpital Cantonal Universitaire de Geneve, Geneva

REFERENCES:
- [Background] Garg S, Serruys P, Onuma Y, Dorange C, Veldhof S, Miquel-Hebert K, Sudhir K, Boland J, Huber K, Garcia E, te Riele JA; SPIRIT II Investigators. 3-year clinical follow-up of the XIENCE V everolimus-eluting coronary stent system in the treatment of patients with de novo coronary artery lesions: the SPIRIT II trial (Clinical Evaluation of the Xience V Everolimus Eluting Coronary Stent System in the Treatment of Patients with de novo Native Coronary Artery Lesions). JACC Cardiovasc Interv. 2009 Dec;2(12):1190-8. doi: 10.1016/j.jcin.2009.10.002. PMID 20129545
- [Result] Serruys PW, Ruygrok P, Neuzner J, Piek JJ, Seth A, Schofer JJ, Richardt G, Wiemer M, Carrie D, Thuesen L, Boone E, Miquel-Herbert K, Daemen J. A randomised comparison of an everolimus-eluting coronary stent with a paclitaxel-eluting coronary stent:the SPIRIT II trial. EuroIntervention. 2006 Nov;2(3):286-94. PMID 19755303
- [Result] Ruygrok PN, Desaga M, Van Den Branden F, Rasmussen K, Suryapranata H, Dorange C, Veldhof S, Serruys PW. One year clinical follow-up of the XIENCE V Everolimus-eluting stent system in the treatment of patients with de novo native coronary artery lesions: the SPIRIT II study. EuroIntervention. 2007 Nov;3(3):315-20. doi: 10.4244/eijv3i3a58. PMID 19737711
- [Result] Khattab AA, Richardt G, Verin V, Kelbaek H, Macaya C, Berland J, Miquel-Hebert K, Dorange C, Serruys PW. Differentiated analysis of an everolimus-eluting stent and a paclitaxel-eluting stent among higher risk subgroups for restenosis: results from the SPIRIT II trial. EuroIntervention. 2008 Mar;3(5):566-73. doi: 10.4244/eijv3i5a102. PMID 19608482
- [Result] Wiemer M, Seth A, Chandra P, Neuzner J, Richardt G, Piek JJ, Desaga M, Macaya C, Bol CJ, Miquel-Hebert K, De Roeck K, Serruys PW. Systemic exposure of everolimus after stent implantation: a pharmacokinetic study. Am Heart J. 2008 Oct;156(4):751.e1-7. doi: 10.1016/j.ahj.2008.07.005. PMID 18926156
- [Result] SPIRIT II study: A clinical evaluation of the XIENCE V everolimus eluting coronary stent system in the treatment of patients with de novo native coronary artery lesions. Serruys Patrick W (Reprint). Erasmus MC, Ctr Thorax, Rotterdam, Netherlands. Journal of the American College of Cardiology 51 ( 10, Suppl. A ): p A261 MAR 11 2008
- [Result] A clinical evaluation of the XIENCE V everolimus eluting coronary stent system in the treatment of patients with cle novo native coronary artery lesions. Ruygrok Peter(Reprint). Auckland City Hosp, Auckland, New Zealand Journal: Journal of the American College of Cardiology 49 ( 9, Suppl. B ): p 28B-29B MAR 6 2007 2007 i2 Summit 2007 on Innovation in Intervention New Orleans, LA, USA March 24 -27, 2007; 20070324 ISSN: 0735-1097
- [Result] A clinical evaluation of the XIENCE V Everolimus Eluting CSS in the treatment of patients with de novo, native coronary artery lesions. Pharmaco kinetic substudy. Seth A (Reprint); Neuzner J; Richardt G; Wiemer M; Piek J J; Desaga M; Macaya C; Serruys P W; Spirit II Investigators (Reprint) Author Address: Max Hosp, Vasc Inst, New Delhi, India. European Heart Journal 27 ( Suppl. 1 ): p 767 AUG 2006 2006 World Congress of Cardiology Barcelona, SPAIN September 02 -06, 2006; 20060902 ISSN: 0195-668X Document Type: Meeting; Meeting Poster
- [Result] Serruys, P. SPIRIT II Study: A Clinical Evaluation of the XIENCE™ V Everolimus Eluting Coronary Stent System in the Treatment of Patients with de novo Native Coronary Artery Lesions. European Society of Cardiology - ESC Congress 2006
- [Result] Serruys, P. SPIRIT II Clinical Study: A clinical evaluation of the XIENCE™ V Everolimus Eluting CSS in the treatment of patients with de novo, native coronary artery lesions - IVUS substudy. Transcatheter Cardiovascular Therapeutics - TCT Congress 2006
- [Result] Claessen BE, Beijk MA, Legrand V, Ruzyllo W, Manari A, Varenne O, Suttorp MJ, Tijssen JG, Miquel-Hebert K, Veldhof S, Henriques JP, Serruys PW, Piek JJ. Two-year clinical, angiographic, and intravascular ultrasound follow-up of the XIENCE V everolimus-eluting stent in the treatment of patients with de novo native coronary artery lesions: the SPIRIT II trial. Circ Cardiovasc Interv. 2009 Aug;2(4):339-47. doi: 10.1161/CIRCINTERVENTIONS.108.831800.108.831800. Epub 2009 Jul 22. PMID 20031737
- [Result] Onuma Y and Serruys P. The SPIRIT II Study - A Clinical Evaluation of the XIENCE V® Everolimus Eluting Coronary Stent System in the Treatment of Patients With De Novo Native Coronary Artery Lesions: 4 Year Clinical Results. American College of Cardiology - ACC '10& i2 Summit 2010.
- [Derived] Genereux P, Rutledge DR, Palmerini T, Caixeta A, Kedhi E, Hermiller JB, Wang J, Krucoff MW, Jones-McMeans J, Sudhir K, Simonton CA, Serruys PW, Stone GW. Stent Thrombosis and Dual Antiplatelet Therapy Interruption With Everolimus-Eluting Stents: Insights From the Xience V Coronary Stent System Trials. Circ Cardiovasc Interv. 2015 May;8(5):e001362. doi: 10.1161/CIRCINTERVENTIONS.114.001362. PMID 25940520
- [Derived] Muramatsu T, Onuma Y, van Geuns RJ, Chevalier B, Patel TM, Seth A, Diletti R, Garcia-Garcia HM, Dorange CC, Veldhof S, Cheong WF, Ozaki Y, Whitbourn R, Bartorelli A, Stone GW, Abizaid A, Serruys PW; ABSORB Cohort B Investigators; ABSORB EXTEND Investigators; SPIRIT FIRST Investigators; SPIRIT II Investigators; SPIRIT III Investigators; SPIRIT IV Investigators. 1-year clinical outcomes of diabetic patients treated with everolimus-eluting bioresorbable vascular scaffolds: a pooled analysis of the ABSORB and the SPIRIT trials. JACC Cardiovasc Interv. 2014 May;7(5):482-93. doi: 10.1016/j.jcin.2014.01.155. Epub 2014 Apr 16. PMID 24746650
- [Derived] Onuma Y, Miquel-Hebert K, Serruys PW; SPIRIT II Investigators. Five-year long-term clinical follow-up of the XIENCE V everolimus-eluting coronary stent system in the treatment of patients with de novo coronary artery disease: the SPIRIT II trial. EuroIntervention. 2013 Jan 22;8(9):1047-51. doi: 10.4244/EIJV8I9A161. PMID 23339811
- [Derived] Claessen BE, Smits PC, Kereiakes DJ, Parise H, Fahy M, Kedhi E, Serruys PW, Lansky AJ, Cristea E, Sudhir K, Sood P, Simonton CA, Stone GW. Impact of lesion length and vessel size on clinical outcomes after percutaneous coronary intervention with everolimus- versus paclitaxel-eluting stents pooled analysis from the SPIRIT (Clinical Evaluation of the XIENCE V Everolimus Eluting Coronary Stent System) and COMPARE (Second-generation everolimus-eluting and paclitaxel-eluting stents in real-life practice) Randomized Trials. JACC Cardiovasc Interv. 2011 Nov;4(11):1209-15. doi: 10.1016/j.jcin.2011.07.016. PMID 22115661
- [Derived] Planer D, Smits PC, Kereiakes DJ, Kedhi E, Fahy M, Xu K, Serruys PW, Stone GW. Comparison of everolimus- and paclitaxel-eluting stents in patients with acute and stable coronary syndromes: pooled results from the SPIRIT (A Clinical Evaluation of the XIENCE V Everolimus Eluting Coronary Stent System) and COMPARE (A Trial of Everolimus-Eluting Stents and Paclitaxel-Eluting Stents for Coronary Revascularization in Daily Practice) Trials. JACC Cardiovasc Interv. 2011 Oct;4(10):1104-15. doi: 10.1016/j.jcin.2011.06.018. PMID 22017936
- [Derived] Caixeta A, Lansky AJ, Serruys PW, Hermiller JB, Ruygrok P, Onuma Y, Gordon P, Yaqub M, Miquel-Hebert K, Veldhof S, Sood P, Su X, Jonnavithula L, Sudhir K, Stone GW; SPIRIT II and III Investigators. Clinical follow-up 3 years after everolimus- and paclitaxel-eluting stents: a pooled analysis from the SPIRIT II (A Clinical Evaluation of the XIENCE V Everolimus Eluting Coronary Stent System in the Treatment of Patients With De Novo Native Coronary Artery Lesions) and SPIRIT III (A Clinical Evaluation of the Investigational Device XIENCE V Everolimus Eluting Coronary Stent System [EECSS] in the Treatment of Subjects With De Novo Native Coronary Artery Lesions) randomized trials. JACC Cardiovasc Interv. 2010 Dec;3(12):1220-8. doi: 10.1016/j.jcin.2010.07.017. PMID 21232715